CLINICAL TRIAL: NCT05296161
Title: Efficacy, Safety and Cost-effectiveness of B Cell Tailored Ocrelizumab Versus Standard Ocrelizumab in Relapsing Remitting Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: B Cell Tailored Ocrelizumab Versus Standard Ocrelizumab in Relapsing Remitting Multiple Sclerosis
Acronym: BLOOMS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Zoé van Kempen, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021.0639
Record Dates: First submitted 2022-02-18; First posted 2022-03-25 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: ocrevus; ocrelizumab; personalised dosing
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled non-inferiority trial in The Netherlands
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard interval dosing (No Intervention): The standard group will receive ocrelizumab every 24 weeks following the current label.
- Personalized B cell tailored ocrelizumab treatment (Experimental): The personalized group will start with B cell measurements 24 weeks after the last infusion (baseline). The infusion interval will never be shorter than 24 weeks. The personalized group will start the study with a possible extension of the interval. The infusion will be postponed as long as CD19 B cell count stays below 10 cells/µL (determined every 4 weeks). When CD19 B cell count exceeds or is equal to 10 cells/µL, ocrelizumab infusion will be scheduled within two weeks
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Personalized B cell tailored ocrelizumab treatment
  Other Names: ocrevus
  Arms: Personalized B cell tailored ocrelizumab treatment

SUMMARY:
Rationale: B-cell depleting therapies like ocrelizumab are very effective in the treatment of relapsing remitting multiple sclerosis (RRMS). As B cell repopulation varies extensively between individuals (ranging from 27-175 weeks), using a treatment scheme with a fixed infusion interval may be suboptimal. So far personalized adapted treatment of ocrelizumab in RRMS has not been studied in a prospective setting.

Objective: Evaluating the efficacy, safety and cost-effectiveness of ocrelizumab when administered in personalized B cell tailored intervals in RRMS patients.

Study design: This is a national multicenter randomized controlled trial with 96 week follow-up.

Study population: The study population consists of 296 adult RRMS patients who have received ocrelizumab treatment for a minimum of 12 months (2x 300 mg infusion and 1x 600mg infusion).

Intervention: Patients will be randomized into the standard interval group (600 mg infusions every 24 weeks) or the personalized interval group in which the infusions will be extended as long as the serum CD19 B cell count is below 10 CD19 cells/µL, determined every 4 weeks.

Main study parameters: To conclude non-inferiority of personalized B cell tailored ocrelizumab there will be two co-primary endpoints: 1. the difference of percentage of confirmed relapse-free patients between the two groups after 96 weeks and 2. the difference of percentage of patients free from new/enlarging T2 lesions on MRI between the two groups after 96 weeks. Secondary study parameters are number of confirmed relapses, annualized relapse rate, number of new T2 lesions and brain atrophy on MRI, disability progression, no evidence of disease activity (NEDA), MS disease biomarkers (serum neurofilament light), quality of life, burden of treatment, immunoglobulin levels and (serious) adverse events including occurrence of infections and COVID-19. Furthermore, various immune cell subsets will be studied in relation to ocrelizumab concentration in a subgroup.

Nature and extent of the burden and risks: All patients will be subjected to visits every 24 weeks including clinical scoring and questionnaires. Blood samples and MRI scans will be taken and performed every 48 weeks. Continuous assessment of key stroke dynamics on the patients smartphone and monthly digital cognitive test and walk test will be performed in most patients. As CD19 B cells are kept near complete depletion, the estimated risk of recurrence of disease activity is very low.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of relapsing remitting multiple sclerosis according to the 2017 McDonald criteria34
* EDSS score of 0 to 6.5
* Treatment with ocrelizumab for a minimum of 48 weeks (two 300 mg infusions and one 600 mg infusion)

Exclusion Criteria:

* Previous treatment with alemtuzumab, cladribine or stem cell transplantation
* Relapse in the past 3 months prior to inclusion
* Subsequent treatment with another DMT next to ocrelizumab in the past 6 months prior to inclusion
* Inability to undergo regular MRI scanning
* Women who are pregnant or expect to become pregnant during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 296 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Confirmed relapse-free patients | 96 weeks
  Difference of percentage of confirmed relapse-free patients between the two treatment groups after 96 weeks follow-up.
Change of T2 lesions on brain MR | 96 weeks
  Difference of percentage of patients without new/enlarging T2 MRI lesions between the two treatment groups after 96 weeks follow-up.

SECONDARY OUTCOMES:
Annualized relapse rate | Baseline, year 1, year 2
  Clinical relapses during B-cell tailored dosing
Total number of active (new and/or enlarging) T2 lesions on brain MRI | Baseline, year 1, year 2
  In comparison to the baseline MRI and number of active MRI scans.
Disability progression during follow-up | Baseline, 6 months,12 months, 18 months, 24 months
  Disability progression measured on the Expanded Disability Status Scale (EDSS)
Disability progression during follow-up | Baseline, year 1, year 2
  Disability progression measured on the Expanded Disability Status Scale (EDSS)
Brain atrophy | Baseline, year 1, year 2
  Rate of brain atrophy comparing baseline MRI and MRI at 96 weeks.
NEDA (no evidence of disease activity) | 96 weeks
  NEDA is defined as absence of confirmed relapses, MRI disease activity (new/enlarging T2 lesions) and confirmed disability progression.
Change of neurofilament light | 96 weeks
  Measured in serum
Change of quality of life | Baseline, year 1, year 2
  Measured by the Multiple Sclerosis Impact Scale (MSIS-29)
Change of burden of treatment | Baseline, year 1, year 2
  measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Ocrelizumab wearing-off effect | Baseline, year 1, year 2
  Presence of a possible wearing-off effect measured by a questionnaire developed by the Amsterdam MS Center
IgG levels | Baseline, year 1, year 2
  Change of IgG levels
Cost analysis | 96 weeks
  Cost-utility analysis using EuroQol 5D (EQ-5D)
Disability progression: decrease of hand mobility | Baseline, 6 months,12 months, 18 months, 24 months
  Significant decrease of hand mobility measured by an app that analyses key stroke dynamics. The dynamics are measured continuously and analysed every 6 months.
Disability progression: two minute walking distance | Baseline, 6 months,12 months, 18 months, 24 months
  Significant decrease of walking distance measured by an app that analyses distance using GPS signal. The test is taken monthly and analysed every 6 months.
Disability progression: cognitive impairment | Baseline, 6 months,12 months, 18 months, 24 months
  Significant decrease of cognitive impairment measured by an app that is validated for a digital Symbol Digit Modalities Test (SDMT). The test is taken monthly and analysed every 6 months.

OTHER OUTCOMES:
Trough ocrelizumab concentration | 24 weeks, 48 weeks, 72 weeks, 96 weeks
  in serum
Intra-individual course and stability B-cell counts and subsets from whole blood | 24 weeks, 48 weeks, 72 weeks, 96 weeks
  In a subgroup of patients cell subsets including CD4+ T cells, CD8+ T cells, CD20+ T cells, CD3-D56+ NK cells, and various B cell subsets (CD19+CD27- naive B cells, CD19+CD27+ memory B cells, CD19+CD27+IgD-IgM- switched memory B cells and CD19+CD27+IgD+ marginal zone B cells) will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Joep Killestein, Prof., Principal Investigator — Amsterdam UMC, location VU
Locations (1):
- Amsterdam UMC, location VU, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After medical ethical commitee approved the study protocol.